CLINICAL TRIAL: NCT05571085
Title: Effects of Core Stabilization and PNF Exercises on Cor Muscle Activation in Obese Children: A Randomized Controlled Study
Brief Title: Core Stabilization and PNF Exercises on Cor Muscle Activation in Obese Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Selma Uzuner, Msc. Physiotherapist, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USelma
Record Dates: First submitted 2022-06-25; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: core muscle activation; Exercise; Core stability; pediatrics
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core Stability Exercises group (Experimental): Core stabilization exercises will be performed based on the program recommended by Jeffrey. Each session will take 40-50 minutes. The program consists of a 5-minute warm-up, 40-minute main exercise and a 5-minute cool-down period.
  Children will be taught the abdominal cupping technique during the first two weeks of the exercises.
  Interventions: Other: Core Stability Exercises
- PNF Exercise Program (Other): PNF exercises will consist of a 5-minute warm-up, 40-minute main exercise and a 5-minute cool-down period, with each session lasting 40-50 minutes.
  Individuals will be taught the abdominal cupping technique during the first two weeks of the program.
  Interventions: Other: PNF Exercise Program
- Control Group (No Intervention): No treatment program was applied. As a result of the study, an effective exercise program will be recommended to the participants.

INTERVENTIONS:
Other: Core Stability Exercises — Core stabilization exercises will be performed based on the program recommended by Jeffrey. Each session will take 40-50 minutes. The program consists of a 5-minute warm-up, 40-minute main exercise and a 5-minute cool-down period.
  Arms: Core Stability Exercises group
Other: PNF Exercise Program — PNF exercises will consist of a 5-minute warm-up, 40-minute main exercise and a 5-minute cool-down period, with each session lasting 40-50 minutes.
  Arms: PNF Exercise Program

SUMMARY:
The aim of this study is to examine the effects of core stabilization and PNF exercises on core muscle activation in obese children.In the study, the initial sample size was calculated as 66 people, under the assumptions that the comparisons between groups would be made with one-way analysis of variance (ANOVA), 3 groups would be included in the study, α= 0.05, β= 0.20 and the effect size would be f= 0.40. The study will be conducted on children between the ages of 10-13 who have a BMI value above the 95% percentile according to age and gender.After recording the sociodemographic information of the individuals, body composition, core muscle activation level, lumbar region muscle endurance, lumbar joint position sense, body image, static and dynamic balances, level of enjoyment of physical activity, physical activity level and pediatric quality of life scale before treatment, 8 weeks of treatment will be measured by the evaluator at the end of the 12-week follow-up period. The level of core muscle activation will be used as the primary outcome measure in the study.

DETAILED DESCRIPTION:
1. Socio-demographic Characteristics: Age, gender, height, body weight, body mass index (BMI) and dominant aspects of individuals will be recorded. The Family Income Scale will be used to evaluate the socio-economic status of the family. The Family Income Scale is a 4-item scale developed by WHO for school-age children as an alternative to measure the level of family welfare. The scale asks children questions about their family, about cars, bedrooms, vacations, and computers.
2. Level of Core Muscle Activation Core muscle strength will be measured using Pressure Biofeedback, a simple and applicable equipment. Children will be asked to perform abdominal cupping via pressure biofeedback. The pressure will then be increased and the child will be advised to maintain constant pressure throughout the test. The level at which the individual maintains a constant pressure for 10 seconds will be noted by the researcher and then these values will be graded according to the Sahrmann
3. Core Stability Test. When the abdominal cupping technique is done correctly, there should be no change in pressure. There are 5 levels in the Sahrmann test. In order to determine the level, the positions specified in order will be applied.
4. Lateral Flexion, Extension and Flexion endurance tests were evaluated with the McGill Core Endurance Test.
5. Joint Position Sense In order to evaluate the joint position sense of the lumbar region, a 10 cm tape measure and a laser pointer placed on the tripod will be used. Participants will be seated on a stool with their feet supported on the floor and their hips and knees flexed to 90 degrees. The distance between the back leg of the stool and the tripod will be 50 cm. A 10 cm tape measure will be placed in the lower lumbar area. The point of the tape measure showing 0 cm will be placed on the sacral 1st segment (S1) and the laser pointer will be positioned on this point. This point will be used as the starting point (neutral position).

   Each participant will be asked to remember and maintain their starting position (neutral position). He will then be asked to move his pelvis from maximum anterior tilt to maximum posterior tilt, hold each position for 5 seconds, and return to the starting position. Then the point of the laser beam falling on the tape measure will be recorded in centimeters. The distance between the starting position (neutral position) and the neutral position of the individual after tilt will be interpreted as an absolute error. Before starting the test, participants will be allowed to practice twice. The test will be repeated 3 times using 1-minute rest intervals and the average value will be used for analysis.
6. Children's Body Image Scale Body image will be measured using the Children's Body Image Scale. There are separate versions of the scale for boys and girls. The scale includes 7 gender-specific images in anatomical position. There are 7 male and 7 female photographs on the scale for each edition. Each photo represents a different BMI range. Pictures are ranked from 1 to 7 according to increase in BMI. BMI values representing men and women are given in the table.

   Children will be asked to mark the picture according to their perceived body size and shape. Calculation will be made by subtracting the number equivalent to the actual BMI value from the detected number. The score range is from -6 to +6, negative scores mean that he perceives himself as smaller than he is, zero indicates the right choice, and positive scores mean that he sees himself as overweight.
7. Balance 7.1 One Leg Standing Test This test, which will be used to evaluate static balance, will be performed on the dominant lower extremity. As a starting position, individuals will be asked to stand on two legs with their hands at the waist and feet shoulder-width apart. With the start command, the time will be started when the individuals bring the other knee to 90 degrees flexion position and stand on their dominant feet. The test will be terminated if the standing foot is not in contact with the ground, the body sway increases, or the above foot touches the ground. At the end of the test, the time on the stopwatch will be recorded in seconds. The test will be repeated three times, with a 60-second rest break between repetitions, and the average of the three results will be calculated. 6.2. "Y" Balance Test The dynamic balance of children will be evaluated with the Y test.
8. Pediatric Quality of Life Scale (PedsQL) PedsQL is a quality of life scale created by Varni et al to measure the health-related quality of life of children and adolescents aged 2-18. Turkish validity and reliability studies were conducted by Memik Nç et al. in 2007 for 13-18 age groups and in 2008 for 8-12 age groups.

   The scale has two different forms, a self-report scale and a parent scale, prepared for the age groups of 2-4, 5-7, 8-12 and 13-18, taking into account the characteristics of the age group. It consists of a total of 23 items and 4 subsections. Physical health consists of emotional, social and school functionality. A raw score between 0-4 is taken for each item. "0"= No problem, "1"= Almost no problem, "2"=Sometimes problem, "3"=Usually problem, "4"=Almost always problem. The raw scores obtained are re-scored to be between 0-100 (0=100, 1=75, 2=50, 3=25.4=0). A higher total score indicates that the individual's quality of life is higher. The sum of the scores obtained from the 8 items in the physical health subscale gives the Physical Health Summary score. The Psychosocial Health Summary Score is determined by the sum of the scores obtained from the Emotional, Social, and School Functioning subscales. If the answers given in the scale are less than 50%, it is not considered as missing data. Missing items are not taken into account and the scale scores are calculated as the sum of the answers divided by the number of items answered in each area. If the answers given in the scale are more than 50%, it is considered as missing data and no scoring is made for that child.
9. Level of Enjoyment of Physical Activity Physical Activity Enjoyment Scale-Short Form will be used to measure the level of enjoyment of physical activity. Physical Activity Enjoyment Scale Moore et al. It has been adapted for use by children and developed as the Physical Activity Enjoyment Scale-Short Form. The scale is a one-dimensional scale with 18 items. Instead of a 7-point Likert-type scale expressing opposite situations in short form, 2 items were removed to make it more understandable for children, and a 5-point Likert-type scale was created by writing more clearly in other items. The scale consists of 5 items to reflect the aims of the study and to determine the enjoyment while continuing the activities in the study.

EDUCATIONAL PROGRAM Individuals will be randomly divided into 3 groups using the minimization program running under the DOS operating system. Minimization will be done by considering age, gender, socioeconomic level and physical activity levels. Core stabilization exercises will be applied to the first group and PNF exercises will be applied to the second group. The third group will be the control group and the individuals in this group will not be interfered with. Exercise programs will be performed as 3 sessions per week for 8 weeks.

Core Stability Exercises:

Core stabilization exercises will be performed based on the program recommended by Jeffrey. Each session will take 40-50 minutes. The program consists of a 5-minute warm-up, 40-minute main exercise and a 5-minute cool-down period.

Children will be taught the abdominal cupping technique during the first two weeks of the exercises. A Pressure Biofeedback device will be used to ensure that children learn correctly. Before starting the contraction, the device will be inflated to a pressure of 40 mmHg and participants will be asked to perform predominantly diaphragmatic breathing. The participant will be asked to stay between these values, as contraction of the transversus abdominus muscle results in a pressure increase ranging from 4-10 mmHg. After the participants learn the abdominal cupping technique, they will move on to core stability exercises. During all exercises, children will be asked to protect their trunks as they have learned in the abdominal cupping technique.

Core stabilization exercises include exercises of increasing difficulty that focus on strengthening the abdominal, low back, and pelvic muscles. Jeffreys' exercise protocol includes 3 levels, starting with level 1 and gradually progressing to level 3. Level 1 consists of static contraction training performed in a stable state. Level 2 includes dynamic training in stable condition and level 3 dynamic and resistance training in unstable condition. Pilates balls will be used to create the unstable condition. Details of the program are presented below.

ELIGIBILITY:
Inclusion Criteria:

* Having a BMI value over the 95% percentile according to age and gender,
* Not included in an ongoing diet program for the last 3 months,
* Children who have not participated in an exercise or sports program for the last 6 months will be included.

Exclusion Criteria:

* Having a chronic disease that requires continuous drug use,
* Having chronic pain that will prevent them from exercising,
* Having a disease of neuromuscular origin,
* Having spinal anomaly,
* Having a history of spinal surgery,
* Children with spinal and sacroiliac joint dysfunction, history of injury or trauma will not be included in the study.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-11-28 (Estimated); Study Completion 2022-12-03 (Estimated)

PRIMARY OUTCOMES:
Core muscle strength | Change from baseline at 8 weeks and 12 weeks after the intervention.
  Core muscle strength will be measured using a simple and feasible equipment, Pressure Biofeedback (Chattanooga Group Inc., Hixson, TN, USA).

SECONDARY OUTCOMES:
McGill Core Endurance Tests | Change from baseline at 8 weeks and 12 weeks after the intervention.
  Children's trunk flexion, extension and lateral flexion endurance will be evaluated.
Joint Position Sense | Change from baseline at 8 weeks and 12 weeks after the intervention.
  Joint Position Sense In order to evaluate the joint position sense of the lumbar region, a 10 cm tape measure and a laser pointer placed on the tripod will be used.
Children's Body Image Scale | change from baseline at 8 weeks and 12 weeks after the intervention
  Body image will be measured using the Children's Body Image Scale. There are separate versions of the scale for boys and girls. The scale includes 7 gender-specific images in anatomical position. There are 7 male and 7 female photographs on the scale for each edition. Each photo represents a different BMI range. Pictures are ranked from 1 to 7 according to increase in BMI. BMI values representing men and women are given in the table.
  Children will be asked to mark the picture according to their perceived body size and shape. Calculation will be made by subtracting the number equivalent to the actual BMI value from the detected number. The score range is from -6 to +6, negative scores mean that he perceives himself as smaller than he is, zero indicates the right choice, and positive scores mean that he sees himself as overweight.
Dynamic Balance test | change from baseline at 8weeks and 12 weeks after the intervention
  Y balance test test will be used for dynamic balance in children.
Static Balance Test | change from baseline at 8weeks and 12 weeks after the intervention
  One leg standing test will be used for static balance in children.
Pediatric Quality of Life Scale (PedsQL) | change from baseline at 8 weeks and 12 weeks after the intervention
  PedsQL is a quality of life scale created by Varni et al. to measure the health-related quality of life of children and adolescents aged 2-18.It consists of a total of 23 items and 4 subsections. Physical health consists of emotional, social and school functionality. A raw score between 0-4 is taken for each item. "0"= No problem, "1"= Almost no problem, "2"=Sometimes problem, "3"=Usually problem, "4"=Almost always problem. The raw scores obtained are re-scored to be between 0-100 (0=100, 1=75, 2=50, 3=25.4=0). A higher total score indicates that the individual's quality of life is higher.
Physical Activity Level | change from baseline at 8 weeks and 12 weeks after the intervention
  The Physical Activity Questionnaire for Older Children (PAQ-C) will be used to determine the physical activity level of children.

CONTACTS AND LOCATIONS:
Overall Officials: SELMA UZUNER, MSc, Principal Investigator — selmauzuner10@gmail.com; EMİNE HANDAN TÜZÜN, PROF, Study Director — selmauzuner10@gmail.com
Locations (1):
- Selma Uzuner, Famagusta, Cyprus